CLINICAL TRIAL: NCT02625727
Title: Comparison of Therapeutic Effects of Hyaluronic Acid vs. Hyaluronic Acid Combined Corticosteroid on Knee Osteoarthritis: A Double Blind, Randomized-controlled Clinical Trial
Brief Title: Effects of Hyaluronic Acid vs. Hyaluronic Acid on Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, associate professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST104-2314-B-341-001
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Physical Activity
Keywords: knee osteoarthritis; hyaluronic acid; corticosteroid; intra-articular injection; therapeutic effect
MeSH Terms: conditions — Motor Activity; Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hyaluronic acid group (Experimental): hyaluronic acid injection
  Interventions: Other: hyaluronic acid
- hyaluronic acid and corticosteroid group (Active Comparator): hyaluronic acid combined corticosteroid injection
  Interventions: Other: hyaluronic acid combined corticosteroid

INTERVENTIONS:
Other: hyaluronic acid — compare the therapeutic effects of hyaluronic acid injection and hyaluronic acid combined corticosteroid injection to patients with knee osteoarthritis
  Arms: hyaluronic acid group
Other: hyaluronic acid combined corticosteroid — compare the therapeutic effects of hyaluronic acid injection and hyaluronic acid combined corticosteroid injection to patients with knee osteoarthritis
  Arms: hyaluronic acid and corticosteroid group

SUMMARY:
Using double blind, randomized controlled design to study the immediate, short-term and intermediate-term therapeutic effects of ultrasound guided hyaluronic acid injection and hyaluronic acid combined corticosteroid injection to patients with knee osteoarthritis.

DETAILED DESCRIPTION:
A total of 76 patients will be collected. The participants will be randomized into two groups, including hyaluronic acid injection group and hyaluronic acid combined corticosteroid injection group.

Physical activity will be evaluated. The hyaluronic acid group will receive three times of hyaluronic acid injection per week in three weeks; the hyaluronic acid combined corticosteroid group will receive hyaluronic acid combined corticosteroid injection in the first week, followed by hyaluronic acid injection at the second and third week.

Re-evaluation will be arranged at after one week of injection, after two weeks of injection, one week after injection, one month after injection, three months after injection, and six month after injection.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of knee with Kellgren/Lawrence grade II or III

Exclusion Criteria:

* Who have implant in knee
* History of neurological deficit, such as stroke

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
physical activity | changes from baseline at after one week of injection, after two weeks of injection, one week after injection, one month after injection, three months after injection, and six month after injection

SECONDARY OUTCOMES:
functional performance (Western Ontario and McMaster Universities Osteoarthritis index) | changes from baseline at after one week of injection, after two weeks of injection, one week after injection, one month after injection, three months after injection, and six month after injection
functional performance (Knee injury and Osteoarthritis Outcome Score) | changes from baseline at after one week of injection, after two weeks of injection, one week after injection, one month after injection, three months after injection, and six month after injection

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — associate professor
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan